CLINICAL TRIAL: NCT04319016
Title: Clinical Characteristics of Coronavirus Disease 2019 (COVID-19) in Pregnancy
Acronym: COVID-preg
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gabriele Saccone, principal investigator, medical doctor, Federico II University
Other Study IDs: 145/20
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Infection Viral
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: pregnant women with laboratory-confirmed 2019-n-CoV — Clinical records and compiled data of all consecutive hospitalized and outpatient pregnant women with laboratory-confirmed 2019-n-CoV were included in a merged database

SUMMARY:
The Novel Coronavirus (2019-nCoV), also known as Wuhan coronavirus, causes the 2019-nCoV acute respiratory disease.

DETAILED DESCRIPTION:
Coronaviruses (CoVs) are the largest group of viruses belonging to the Nidovirales order. They are enveloped, non-segmented positive-sense RNA viruses.

Coronavirus are believed to cause a significant proportion of all common colds in adults and children. The Novel Coronavirus (2019-nCoV), also known as Wuhan coronavirus, causes the 2019-nCoV acute respiratory disease. The initial cases of 2019-nCoV occurred in Wuahn, China in December 2019.

A recent review evaluated the potential impact of 2019-nCoV in pregnancy. The authors reported published data on CoVs in pregnant women, including 2019-nCoV, severe acute respiratory syndrome (SARS-COV) and Middle East respiratory syndrome (MERS-COV). The review included 12 women with SARS-COV,4 11 women MERS-COV,5 and 9 women with 2019-n-CoV6 in pregnancy. No cases of vertical trasmission were reported, but the authors showed an high rate of preterm birth (45.8%), cesarean delivery (70.8%), maternal admission to intensive care unit (ICU) (63.3%), and maternal death (18.8%).

The aim of this study was to evaluate the pregnancy and perinatal outcomes of pregnant women with 2019-n-CoV.

This was a multicenter, retrospective, cohort study. Clinical records and compiled data of all consecutive hospitalized and outpatient pregnant women with laboratory-confirmed 2019-n-CoV Data on recent exposure history, clinical symptoms or signs, laboratory findings, and maternal and perinatal outcomes were collected. All medical recors were sent to the coordinator center. Data were entered into a computerized database and cross-checked. If the core data were missing, requests for clarification were sent to the coordinators.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with laboratory-confirmed 2019-n-CoV

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — pregnant women
Study Population: pregnant women with laboratory-confirmed 2019-n-CoV
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Maternal and perinatal outcomes | at the time of delivery
  different maternal and perinatal outcomes were evaluated including: admission to ICU, use of mechanical ventilation, maternal death, early pregnany loss, perinatal death, intrauterine growth restriction (IUGR), preterm birth, mode of delivery, LBW, admission to neonatal ICU (NICU), and clinical or serologic evidence of vertical trasmission

CONTACTS AND LOCATIONS:
Locations (1):
- Gabriele Saccone, Napoli, Italy

IPD SHARING:
Plan to Share IPD: Undecided
not planned yet